CLINICAL TRIAL: NCT06834789
Title: A Phase 1 Study to Evaluate the Safety and Efficacy of Co-administration of AGN-151586 and BOTOX® in Subjects for Treatment of Glabellar Lines (GL)
Brief Title: A Study to Assess the Adverse Events of Intramuscular Injections of AGN-151586 and OnabotulinumtoxinA in Adult Participants for the Change of Glabellar Lines (GL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M25-207
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Glabellar Lines
Keywords: Glabellar Lines; AGN-151586; OnabotulinumtoxinA
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1: AGN-151586 Dose A and OnabotulinumtoxinA (Experimental): Participants will receive a single treatment of AGN-151586 Dose A and OnabotulinumtoxinA.
  Interventions: Drug: AGN-151586; Drug: OnabotulinumtoxinA
- Cohort 2: AGN-151586 Dose B and OnabotulinumtoxinA (Experimental): Participants will receive a single treatment of AGN-151586 Dose B and OnabotulinumtoxinA.
  Interventions: Drug: AGN-151586; Drug: OnabotulinumtoxinA
- Cohort 3: AGN-151586 Dose A and OnabotulinumtoxinA (Experimental): Participants will receive a single treatment of AGN-151586 Dose A and OnabotulinumtoxinA.
  Interventions: Drug: AGN-151586; Drug: OnabotulinumtoxinA
- Cohort 3: AGN-151586 Dose B and OnabotulinumtoxinA (Experimental): Participants will receive a single treatment of AGN-151586 Dose B and OnabotulinumtoxinA.
  Interventions: Drug: AGN-151586; Drug: OnabotulinumtoxinA
- Cohort 3: Placebo and OnabotulinumtoxinA (Experimental): Participants will receive a single treatment of Placebo and OnabotulinumtoxinA.
  Interventions: Drug: OnabotulinumtoxinA; Drug: Placebo

INTERVENTIONS:
Drug: AGN-151586 — Intramuscular injection
  Arms: Cohort 1: AGN-151586 Dose A and OnabotulinumtoxinA; Cohort 2: AGN-151586 Dose B and OnabotulinumtoxinA; Cohort 3: AGN-151586 Dose A and OnabotulinumtoxinA; Cohort 3: AGN-151586 Dose B and OnabotulinumtoxinA
Drug: OnabotulinumtoxinA — Intramuscular injection
Drug: Placebo — Intramuscular injection
  Arms: Cohort 3: Placebo and OnabotulinumtoxinA

SUMMARY:
The objective of this Phase 1 study is to assess the safety and efficacy of single treatment of AGN-151586 and of OnabotulinumtoxinA in the glabellar complex of participants with moderate to severe glabellar lines (GL).

ELIGIBILITY:
Inclusion Criteria:

* Has moderate or severe glabellar lines (GL) at maximum frown as assessed by both the investigator and participant using the Facial Wrinkle Scale (FWS).
* Must be in good health as per investigator's judgment based on medical history, physical examination, vital sign measurements, 12-lead ECG parameters, clinical laboratory evaluations, and neurological assessment.

Exclusion Criteria:

* Active infection or dermatological condition at the treatment injection sites.
* History of immunization to any botulinum neurotoxin serotype or hypersensitivity to any botulinum neurotoxin serotype or any other constituents of the study drug or its excipients, and/or other products in the same class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 10.4 months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Number of Participants with the Presence of Binding and Neutralizing Antidrug Antibodies to AGN-151586 and/or OnabotulinumtoxinA | Up to approximately 10.4 months
  Samples collected from participants treated with AGN-151586 and OnabotulinumtoxinA will be analyzed for antibodies against both AGN-151586 and OnabotulinumtoxinA.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- United States (8):
  - Investigate MD /ID# 270771, Scottsdale, Arizona
  - Eye Research Foundation /ID# 270827, Newport Beach, California
  - Marcus Facial Plastic Surgery /ID# 270770, Redondo Beach, California
  - Skin Research Institute LLC /ID# 270831, Coral Gables, Florida
  - Skincare Physicians /ID# 271018, Chestnut Hill, Massachusetts
  - Wilmington Dermatology Center /ID# 270828, Wilmington, North Carolina
  - Austin Institute for Clinical Research - Pflugerville /ID# 270834, Pflugerville, Texas
  - SkinDC /ID# 270932, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-207